CLINICAL TRIAL: NCT00196651
Title: Randomized Study on HIV Immune and Virological Responses Following the Administration of IL-2 Either Alone or Combined to ALVAC-HIV 1433 and HIV Lipopeptides (LIPO-6T) in Patients Treated Early With HAART During Primary Infection. ANRS 095 PRIMOVAC
Brief Title: HIV Immune and Virological Responses Following the Administration of IL-2 Either Alone or Combined to ALVAC-HIV 1433 and HIV Lipopeptides in Patients Treated Early With HAART During Primary Infection
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Collaborators: Aventis Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANRS 095 PRIMOVAC
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2005-09-20 (Estimated); Status verified 2005-09

CONDITIONS: HIV Infection
Keywords: HIV infection; AIDS Vaccines; ALVAC vaccine; Interleukin-2; Antiretroviral Therapy, Highly Active
MeSH Terms: conditions — HIV Infections | interventions — Interleukin-2; HIV-LIPO-6T

INTERVENTIONS:
Drug: IL-2
Biological: LIPO-6T
Biological: ALVAC VIH 1433

SUMMARY:
HIV-specific immune responses are preserved in patients treated early during primary infection.The trial evaluated whether the addition to HAART of IL-2 alone or combined with an immunization procedure might enhance HIV immune responses and improve viral control after HAART discontinuation

DETAILED DESCRIPTION:
HIV-specific immune responses are preserved in patients treated early during primary infection. The trial evaluated whether the addition to HAART of IL-2 alone or combined with an immunization procedure might enhance HIV immune responses and improve viral control after HAART discontinuation.Patients treated with HAART are randomized to 3 arms:arm1 HAART alone; arm2 with 5 cycles of IL-2 at wk0 ,8 ,16 ,24 and 32;arm3 4 injections of Alvac-HIV 1433 and LIPO-6T at wk0,4,8 followed by 3 cycles of IL-2 at w 16, 24 and 32. HAART is stopped at wk 40 in patient with undetectable plasma viral load. Viral loads and HIV-specific responses are monitored during the therapeutic period and after HAART interruption until w52. HAARTis rei-initiated with viral failure.

ELIGIBILITY:
Inclusion Criteria:

* History of symptomatic HIV primary infection with p24 positive or incomplete Western Blot
* Treatment beginning before 4W after the first primary infection serology
* HAART with IP or NNRTI since one year, wtih no change since 3 months
* Viral load below 50 cp since 6 months
* PN over 1000/mm3;Hb over 10.5g/l;Platelets over 75000/mm3, creatinine below 1.5N; transaminases below 2.5N

Exclusion Criteria:

* Vaccination or chemotherapy or corticosteroid since 3 months
* Evolutive cancer
* pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2000-08; Study Completion 2004-02

PRIMARY OUTCOMES:
Evolution of CD4-CD8 non specific and HIV specific cells, vaccinal peptids and viral load with DNA proviral at W36

SECONDARY OUTCOMES:
Safety of IL-2, ALVAC and LIPO-6T
Tolerability of HAART
Kinetic of viral load rebound with frequency and delay of cv over 10 000 cp and 50 000 cp
Evolution on immune response and predictive value of immunologic parameters on viral load

CONTACTS AND LOCATIONS:
Overall Officials: Cecile Goujard, MD, Principal Investigator — Hopital Kremlin Bicetre Bicetre France; Jean Pierre Aboulker, MD, Study Director — Inserm SC10 France

REFERENCES:
- [Derived] Goujard C, Marcellin F, Hendel-Chavez H, Burgard M, Meiffredy V, Venet A, Rouzioux C, Taoufik Y, El Habib R, Beumont-Mauviel M, Aboulker JP, Levy Y, Delfraissy JF; PRIMOVAC-ANRS 095 Study Group. Interruption of antiretroviral therapy initiated during primary HIV-1 infection: impact of a therapeutic vaccination strategy combined with interleukin (IL)-2 compared with IL-2 alone in the ANRS 095 Randomized Study. AIDS Res Hum Retroviruses. 2007 Sep;23(9):1105-13. doi: 10.1089/aid.2007.0047. PMID 17919105